CLINICAL TRIAL: NCT06019585
Title: Inmobilization With Compression Bandage vs Antebraquial Splint in Distal Radius Fractures Operated by Internal Fixation With Volar Locking Plate: A Pilot Study
Brief Title: Inmobilization With Compression Bandage vs Antebraquial Splint in Distal Radius Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Costa del Sol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 003may21PIInmovilizacionfxd
Record Dates: First submitted 2023-07-24; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Distal Radius Fractures; Internal Fixation; Complications, Mechanical
Keywords: distal radius fractures; volar plate; internal fixation; Inmobilization
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: 2 parallel groups, each one receives one treatment
Who Masked: Outcomes Assessor
Masking Description: Patient receive the correspondant treatment based on the order of an aleatory numbers table
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Splint inmmobilization (Active Comparator): Distal radius fractures fixed with volar locking plate and immobilized with an antebrachial splint for 3 weeks
  Interventions: Device: Splint inmmobilization
- Bandage immovilization (Active Comparator): Distal radius fractures fixed with volar locking plate and immobilized with a compressive bandage for 3 weeks
  Interventions: Device: Bandage immovilization

INTERVENTIONS:
Device: Splint inmmobilization — After internal fixation with volar locking plate, groups of distal radius fractures are inmobilized with a plaster splint of París for 3 weeks
  Arms: Splint inmmobilization
Device: Bandage immovilization — After internal fixation with volar locking plate, groups of distal radius fractures are inmobilized with compressive bandage for 3 weeks
  Arms: Bandage immovilization

SUMMARY:
The aim of this study is to compare functional and radiological results in two groups of distal radius fractures treated with internal fixation with locking plate, and immobilized with antebrachial splint or compression bandage for 3 weeks.

DETAILED DESCRIPTION:
The aim of the study is to compare functional and radiological results as well as to evaluate possible complications in distal radius fractures operated by open reduction and internal fixation with volar locking plate in two groups , one treated with immobilization using a forearm cast for 3 weeks and the other with immobilization using a compression bandage for 3 weeks, based on the hypothesis that compression bandage group could obtain better results in the short term, and none of the treatments is superior to the other after 3 or 6 months of evolution, as indicated by some reviewed studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type A, B, C fractures of AO classification of distal radius fractures
* Patents aged between 18 and 75 years,
* Patients operated on in the first 3 weeks after the trauma, and independent for the basic activities of daily living

Exclusion Criteria:

* Patients with open fractures
* Patients with mental disorders (dementia, alcoholism, etc.),
* Patient dependent for basic activities of daily living
* Patients with fractures with severe articular and metaphyseal comminution and/or severe soft tissue injuries (type 2R3C3 AO),
* Patients with previous diseases or anatomical alterations in the injured wrist (previous fractures, rheumatoid arthritis, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain in Visual Analogue Scale. | 1 year
  Points from 1 to 10. Higher score: worse value. Lower score: better value.
Function in Patient Rated Wrist Evaluation Scale. | 1 year
  Points from 1 to 100. Higher score: worse value. Lower score: better value.
Range Of Motion in Flexion. | 1 year
  Grades from 0 to 70. Higher score: better value. Lower score: worse value.
Range Of Motion in Flexion. | 1 year
  Grades from 0 to 80. Higher score: better value. Lower score: worse value.

SECONDARY OUTCOMES:
Function in Disabilities of Arm, Shoulder and Hand Scale. | 1 year
  Points from 1 to 150. Higher score: worse value. Lower score: better value
Function in Mayo Wrist Score Scale. | 1 year
  Points from 1 to 100. Higher score: worse value. Lower score: better value.
Range of motion in Supination. | 1 year
  Grades from 0 to 90. Higher score: better value. Lower score: worse value.
Number of participants with posoperative complications. | 1 year
  Number of participants per group that suffer some complication or side effect during the follow-up period. Higher number of complications: worse value.
Number of posoperative Fisiotherapy sessions performed. | 1 year
  Number of sessions per participant from 1 to 100. Higher score: worse value. Lower score: better value.
Time of fracture union in radiographs. | 12 weeks
  Number of Weeks from 1 to 12. Higher score: worse value. Lower score: better value.
Number of Instability distal radius fracture Criteria per participant. | 1 year
  Number of criteria from 1 to 6. Higher score: worse value. Lower score: better value.
Grades of Dorsal Displacement in fracture. | 6 weeks
  Grades from -10 to 30 grades. Higher score: worse value. Lower score: better value.
Range of motion in Pronation. | 1 year
  Grades from 0 to 90. Higher score: better value. Lower score: worse value.
Range of motion in Radial Deviation | 1 year
  Grades from 0 to 15. Higher score: better value. Lower score: worse value.
Range of motion in Ulnar deviation. | 1 year
  Grades from 0 to 30. Higher score: better value. Lower score: worse value.
Number of shortening millimeters in fracture. | 6 weeks
  Number of millimeters from 0-10. Higher score: worse value. Lower score: better value.
Number of ulnar variance millimeters in fracture. | 6 weeks
  Number of millimeters from -2 to +4. Higher score: worse value. Lower score: better value.
Number of step-off millimeters in fracture. | 6 weeks
  Number of millimeters from 0 to 4 mm. Higher score: worse value. Lower score: better value.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Izquierdo Fernández, Phd, Study Director — Hospital Reina Sofía ( Córdoba, Spain)
Locations (2):
- Spain (2):
  - Hospital Reina Sofía, Córdoba
  - Hospital Costa del Sol, Málaga

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Delft EAKV, Gelder TGV, Vries R, Vermeulen J, Bloemers FW. Duration of Cast Immobilization in Distal Radial Fractures: A Systematic Review. J Wrist Surg. 2019 Oct;8(5):430-438. doi: 10.1055/s-0039-1683433. Epub 2019 Mar 18. PMID 31579555
- [Result] Quadlbauer S, Pezzei C, Jurkowitsch J, Kolmayr B, Keuchel T, Simon D, Hausner T, Leixnering M. Early Rehabilitation of Distal Radius Fractures Stabilized by Volar Locking Plate: A Prospective Randomized Pilot Study. J Wrist Surg. 2017 May;6(2):102-112. doi: 10.1055/s-0036-1587317. Epub 2016 Aug 5. PMID 28428911
- [Result] Toemen A, Collocott S, Heiss-Dunlop W. Short Term Outcomes Following Open Reduction Internal Fixation Surgery for a Distal Radius Fracture: 2 Week Versus 4 Week Immobilization. A Retrospective Analysis. Geriatr Orthop Surg Rehabil. 2021 Mar 25;12:21514593211004528. doi: 10.1177/21514593211004528. eCollection 2021. PMID 35186419
- [Result] Klein SM, Prantl L, Koller M, Vykoukal J, Dolderer JH, Graf S, Nerlich M, Loibl M, Geis S. Evidence based postoperative treatment of distal radius fractures following internal locking plate fixation. Acta Chir Orthop Traumatol Cech. 2015;82(1):33-40. PMID 25748659
- [Result] Lichtman DM, Bindra RR, Boyer MI, Putnam MD, Ring D, Slutsky DJ, Taras JS, Watters WC 3rd, Goldberg MJ, Keith M, Turkelson CM, Wies JL, Haralson RH 3rd, Boyer KM, Hitchcock K, Raymond L; American Academy of Orthopaedic Surgeons. American Academy of Orthopaedic Surgeons clinical practice guideline on: the treatment of distal radius fractures. J Bone Joint Surg Am. 2011 Apr 20;93(8):775-8. doi: 10.2106/JBJS.938ebo. No abstract available. PMID 21508285
- [Result] Valdes K, Naughton N, Michlovitz S. Therapist supervised clinic-based therapy versus instruction in a home program following distal radius fracture: a systematic review. J Hand Ther. 2014 Jul-Sep;27(3):165-73; quiz 174. doi: 10.1016/j.jht.2013.12.010. Epub 2014 Jan 3. PMID 24508093
- [Result] Driessens S, Diserens-Chew T, Burton C, Lassig E, Hartley C, McPhail S. A retrospective cohort investigation of active range of motion within one week of open reduction and internal fixation of distal radius fractures. J Hand Ther. 2013 Jul-Sep;26(3):225-30; quiz 231. doi: 10.1016/j.jht.2013.05.002. Epub 2013 Jun 14. PMID 23770202
- [Result] Koval K, Haidukewych GJ, Service B, Zirgibel BJ. Controversies in the management of distal radius fractures. J Am Acad Orthop Surg. 2014 Sep;22(9):566-75. doi: 10.5435/JAAOS-22-09-566. PMID 25157038
- [Result] Lozano-Calderon SA, Souer S, Mudgal C, Jupiter JB, Ring D. Wrist mobilization following volar plate fixation of fractures of the distal part of the radius. J Bone Joint Surg Am. 2008 Jun;90(6):1297-304. doi: 10.2106/JBJS.G.01368. PMID 18519324
- [Result] Meinberg EG, Agel J, Roberts CS, Karam MD, Kellam JF. Fracture and Dislocation Classification Compendium-2018. J Orthop Trauma. 2018 Jan;32 Suppl 1:S1-S170. doi: 10.1097/BOT.0000000000001063. No abstract available. PMID 29256945